CLINICAL TRIAL: NCT03196232
Title: Phase 2 Study of Epacadostat (INCB024360) With Pembrolizumab (MK3475) in Metastatic or Unresectable Gastroesophageal Junction and Gastric Adenocarcinoma Requiring Paired Biopsies
Brief Title: Epacadostat and Pembrolizumab in Treating Patients With Metastatic or Unresectable Gastroesophageal Junction or Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: George Albert Fisher (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, George Albert Fisher, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-40823; NCI-2017-00895 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GI0015 (Other: OnCore)
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2020-06-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Recurrent Esophageal Carcinoma; Recurrent Gastric Carcinoma; Stage IV Esophageal Cancer AJCC v7; Stage IV Gastric Cancer AJCC v7; Unresectable Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — epacadostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (epacadostat, pembrolizumab) (Experimental): Participants receive oral epacadostat BID on Days 1 to 21 and pembrolizumab IV over 30 minutes on Day 1, with cycles repeating every 21 days for up to 24 months, in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Epacadostat — Given PO
  Other Names: INCB 024360; INCB024360
Drug: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase 2 trial evaluates the benefit of epacadostat plus pembrolizumab in combination to treat patients with gastroesophageal junction or gastric cancer that has spread to other parts of the body and cannot be removed by surgery. Epacadostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as pembrolizumab, may block tumor growth in different ways by targeting certain cells. Giving epacadostat and pembrolizumab may work better in treating patients with gastroesophageal junction or gastric cancer.

DETAILED DESCRIPTION:
Patients receive epacadostat orally (PO) twice daily (BID) on Days 1 to 21 and pembrolizumab intravenously (IV) over 30 minutes on Day 1. Courses repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 9 weeks for 18 months, and then every 12 weeks thereafter.

PRIMARY OBJECTIVES:

Assess 6-month progression free survival (PFS).

SECONDARY OBJECTIVES:

* To evaluate objective response rate (RR) by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 and immune-related response criteria (irRC).
* Evaluate overall survival (OS).
* Assess the safety and tolerability of epacadostat in combination with pembrolizumab by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03.

TERTIARY OBJECTIVES:

* Determine the responder rate defined as the proportion of subjects with an increased ratio of CD8+ to Treg cells in on-treatment compared with pre-treatment biopsies.
* Identify putative immunologic biomarkers of tumor response.

ELIGIBILITY:
INCLUSION CRITERIA

* ≥ 18 years of age on day of consent
* Histologically-or cytologically-confirmed adenocarcinoma of the distal esophagus [within 5 centimeters of the gastroesophageal junction (GEJ)], gastroesophageal junction or stomach, including HER2+ disease
* Metastatic or unresectable disease, including those with HER2+ disease
* Progressed on at least 1 line of prior therapy for metastatic disease, or intolerant to that therapy if not progressed
* If HER2+ disease, should have received prior trastuzumab
* Life expectancy ≥ 12 weeks
* Eastern Cooperative Oncology (ECOG) Performance Status 0 or 1
* Measurable disease per RECIST v1.1, assessed within 4 weeks prior to study entry
* Tumor deemed amenable to biopsy by core for metastatic site or endoscopic biopsy for primary tumor (for both before and on-treatment biopsies)
* Able to swallow pills
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 3 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception starting with the date of consent through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the date of consent through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Prior authorization by Merck in order to enroll in this study is required if previously treated on any Merck-sponsored pembrolizumab-containing gastric cancer pivotal trial
* Willing to undergo 2 biopsies (before and on-treatment), provided the procedure is not deemed high-risk and is clinically feasible
* Willing and able to provide written informed consent/assent

EXCLUSION CRITERIA

* Known additional malignancy that has progressed or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. EXCEPTION: subjects with previously-treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability. Patients with prior CNS metastases treated with prior radiation therapy (RT) will also need ALL of the following:

  * 2 months off RT before starting study or 4 weeks following radiation therapy (XRT) if magnetic resonance imaging (MRI) is stable and the patient is off steroids
  * Baseline MRI with no edema
  * Stable for at least 8 weeks
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Use of systemic corticosteroids
* Currently, or within 4 weeks of the first planned dose of treatment, receiving an investigational agent and using an investigational device
* Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1, or anyone has not recovered from adverse events (ie, to baseline or ≤ grade 1) due to agents administered more than 4 weeks earlier (EXCEPTION: denosumab for bone metastases is allowed)
* Prior chemotherapy; targeted small molecule therapy; or radiation therapy within 2 weeks prior to study day 1 or who has not recovered from adverse events (ie, to baseline or ≤ grade 1) due to a previously administered agent (EXCEPTION: ≤ grade 2 neuropathy). Recovery from major surgery must be considered adequate prior to starting therapy.
* Prior therapy with indoleamine-pyrrole 2,3-dioxygenase (IDO)-inhibitors
* Prior therapy with monoamine oxidase inhibitors within 21 days before screening
* Presence of a gastrointestinal condition that may affect drug absorption
* Active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents; corticosteroids; or immunosuppressive drugs). EXCEPTION: replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered systemic treatment
* Known hypersensitivity to pembrolizumab and/or epacadostat or any of their excipients
* Known allergy or reaction to any component of either study drug or formulation components
* Received a live vaccine, including live attenuated vaccines (eg, Flu-Mist), within 30 days of planned start of study therapy. EXCEPTION: inactivated flu vaccines such as seasonal influenza vaccines for injection are allowed
* Known active hepatitis B (eg, hepatitis B surface antigen [HBsAg] reactive)
* Known active hepatitis C (eg, hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] detected)
* Known history of active tuberculosis (Bacillus tuberculosis)
* Known history of human immunodeficiency virus (HIV) (HIV 1-2 antibodies)
* Known history of, or any evidence of active, non-infectious pneumonitis
* History of serotonin syndrome after receiving 1 or more serotonergic drugs
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* History or presence of an abnormal electrocardiogram (ECG) which, in the investigator's opinion, is clinically significant
* Corrected QT Fredericia's formula (QTcF) ≥ 480 ms or presence of a left bundle branch block (LBBB); if the QRS duration > 120ms, the JTc can be used in place of the QTcF; the JTc must be < 340 ms
* Active infection requiring systemic therapy
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with pre-screening or screening visit through 120 days after the last dose of study treatment
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A Fisher, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was assessed as the number of participants remaining alive without progression 6 months after beginning treatment. The outcome is reported as a number without dispersion.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Response Rate
Description: Therapeutic response was assessed per the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). Criteria are:
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
  The outcome is reported as the number of participants with a documented clinical response (ie, either PR or CR) at 6 months after initiation of treatment.
Time Frame: Up to 6 months
Population: Not all subjects completed 6 months of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 1
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Overall Response (OR) | 0
  Progressive disease (PD) | 1
  Stable disease (SD) | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was assessed as the number of participants remaining alive 6 months after beginning treatment. The outcome is reported as a number without dispersion.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 3
Participants | 1

4. Secondary Outcome: Number of Adverse Events
Description: Participants were monitored for adverse events. The outcome is reported as the overall number of adverse events of any grade, a number without dispersion.
Time Frame: Up to 6 months
Measure: Number; unit: Adverse events
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 3
Adverse events | 42

5. Secondary Outcome: Number of Adverse Events ≥ Grade 3
Description: Adverse events were assessed per the Common Terminology Criteria for Adverse Events v4.03. The outcome is reported as the number of adverse events ≥ Grade 3, a number without dispersion.
Time Frame: Up to 6 months
Measure: Number; unit: Adverse events
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 3
Adverse events | 2

6. Secondary Outcome: Treatment Delay or Reduction
Description: The assessment for clinical value of the treatment combination included treatment delays or reductions, a measure of how well the combination treatment was tolerated. The outcome is reported as the number of participants that experienced a treatment delay, or reduction in treatment dose level, a number without dispersion.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events reported through 30 days after treatment. Overall mortality was monitored though 6 months.
Arm/Group | Treatment (Epacadostat, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Epacadostat, Pembrolizumab) (N=3)
Jejunal perforation (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Epacadostat, Pembrolizumab) (N=3)
Vomiting (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Jejunal Perforation (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
Sepsis (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Weight Loss (Gastrointestinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Gastrointestinal disorders) | 1 (1)
Cholesterol high (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Gastrointestinal disorders) | 1 (1)
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hair Color Change (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT03196232/Prot_SAP_000.pdf